CLINICAL TRIAL: NCT03722862
Title: Sunfiber and the Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY99994204
Record Dates: First submitted 2018-08-29; First posted 2018-10-29 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Diet Modification

STUDY DESIGN:
Intervention Model Description: 3 arm crossover, randomized
Who Masked: Participant, Investigator
Masking Description: fiber is provided in pouches; coded to treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm (Placebo Comparator): Healthy volunteers will continue normal healthy diet with a placebo.
  Interventions: Dietary Supplement: Placebo
- Low fiber (Experimental): Healthy volunteers will be randomized to receive 3 grams of Sunfiber.
  Interventions: Dietary Supplement: Low fiber
- High fiber (Experimental): Healthy volunteers will be randomized to receive 6 grams of Sunfiber.
  Interventions: Dietary Supplement: High fiber

INTERVENTIONS:
Dietary Supplement: Low fiber — Partially hydrolyzed guar gum (PHGG) commercially available as Sunfiber in 3 gram doses
  Arms: Low fiber
Dietary Supplement: Placebo — Participants will receive the placebo/dextrose.
  Arms: Control Arm
Dietary Supplement: High fiber — Partially hydrolyzed guar gum (PHGG) commercially available as Sunfiber in 6 gram doses
  Arms: High fiber

SUMMARY:
The aim of this study is to look at the effect Sunfiber has on the gut microbiota.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled crossover study with a 2 week washout period. Healthy volunteers will receive placebo, 4 grams, or 8 grams of Sunfiber in addition to their regular diet. Fecal samples will be collected for measurement of bowl function, including the gut microbiota.

ELIGIBILITY:
Inclusion Criteria

* Healthy male or female between the ages of 20-49 years
* Subject has a body mass index of ≥18.5 and ≤30 kg/m2 at screening visit.
* Subject is willing to stick to their normal habitual diet excluding the consumption of any unusual high energy-rich or fat-rich meals or prolonged fasting, etc. through the study period.
* Subject is willing to maintain their habitual physical activity patterns throughout the study period.
* Subject has been weight stable within the last 6 months.
* Subject has no health conditions that would prevent him or her from fulfilling the study requirements as judged by the investigator on the basis of medical history and routine laboratory test results.
* Low fiber consumer (≤14 g per day)
* Subject is willing to follow study procedures and dietary restrictions (ex: stick to habitual diet, refrain from consuming alcohol 24 hours prior to test days).
* Subject understands study procedures and signs forms providing informed consent to participate in the study.

Exclusion Criteria:

* History of a gastrointestinal disorder
* Lactose intolerant
* High fiber consumer (≥15 g per day)
* Use of pre-and probiotics in the past 90 days
* High protein consumer (i.e. vegetarians or those who follow diets high in protein such as paleo)
* History of psychological illness or conditions that may interfere with subjects ability to understand study directions
* Use of antibiotics or signs of active systemic infection in the last 6 months. Subjects who are on hypo/hypercaloric diet aiming for weight loss or weight gain
* History or presence of cancer in the prior 2 years (except for non-melanoma skin cancer).

Currently pregnant, lactating or planning to be pregnant during the study period

* Regular use of dietary supplements (ex: fish oil, riboflavin, etc.), 90 days prior to study inclusion
* Exposure to any non-registered drug product within the last 30 days prior to screening visit
* History of or strong potential for alcohol or substance abuse (within 12 months of screening visit). Alcohol abuse is defined as >60g (men)/40g (women) pure alcohol per day (1.5 L/ 1 l beer resp. 0.75l/0.5l wine).

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-09-14 (Actual)

PRIMARY OUTCOMES:
Analysis of Microbiota | Day 10
  Bacterial phyla, genera, and species of bacteria will be detected using real tijme PCR. All abundances will be calculated and presented as relative levels (relative to the total amount of eubacteriausing a universal eubacteria prijer set)

SECONDARY OUTCOMES:
salivary cortisol | Day 10
  Salivary cortisol will be measured using a competitive immunoassay. 25 ul of saliva will be used in each replicate and results will be compared to a standard curve and calculated as ug/dl.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Food Science and Nutrition, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No